CLINICAL TRIAL: NCT06926582
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Phase II Study to Evaluate Clinical Efficacy and Safety of HS-10374 in Adult Patients With Mild-to-moderate Plaque Psoriasis
Brief Title: A Study to Evaluate Efficacy and Safety of HS-10374 for Mild-to-moderate Plaque Psoriasis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-10374-205
Record Dates: First submitted 2025-04-10; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HS-10374 Dose 1 (Experimental)
  Interventions: Drug: HS-10374 6mg tablets; Drug: HS-10374-matched placebo tablets
- HS-10374 Dose 2 (Experimental)
  Interventions: Drug: HS-10374 6mg tablets
- Placebo (Placebo Comparator)
  Interventions: Drug: HS-10374-matched placebo tablets

INTERVENTIONS:
Drug: HS-10374 6mg tablets — Administered orally QD for 12 weeks
  Arms: HS-10374 Dose 1; HS-10374 Dose 2
Drug: HS-10374-matched placebo tablets — Administered orally QD for 12 weeks
  Arms: HS-10374 Dose 1; Placebo

SUMMARY:
This study has been designed to explore the clinical efficacy and safety of HS-10374 in the treatment of mild-to-moderate plaque psoriasis.

DETAILED DESCRIPTION:
This is a 12-week, multi-center, randomized, double-blind, placebo-controlled, Phase II study. The study duration includes a 4-week screening period, a 12-week placebo-controlled treatment period, and a 4-week follow-up period. All eligible subjects will be randomly assigned in a 2:2:1 ratio to receive HS-10374 Dose 1, HS-10374 Dose 2, or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between the ages of 18-70 years
2. Diagnosis of plaque psoriasis for at least 6 months
3. sPGA score of 2-3, BSA 2-15%, PASI score 2-15
4. Subject must be inadequately controlled with, or intolerant of at least one topical therapy

Exclusion Criteria:

1. Diagnosis of non-plaque psoriasis or drug-induced psoriasis
2. Recent history of infection, history or risk of serious infection
3. Any major illness or evidence of unstable condition of major organ systems including psychiatric disease
4. Any condition possibly affecting the PK process of the study drug
5. Evidence of other skin conditions that would interfere with the evaluation of psoriasis
6. History of hypersensitivity to the ingredients of study drugs, history of anaphylaxis
7. Prior exposure to TYK2 inhibitors
8. Have received the prohibited treatment during the protocol required washout period
9. Any significant laboratory or procedure abnormalities that might place the subject at unacceptable risk during this study period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Estimated)
Dates: Start 2025-04-09 (Estimated); Primary Completion 2026-07-09 (Estimated); Study Completion 2026-12-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving sPGA 0/1 with at least 2 points improvement from baseline at Week 12 | Baseline to Week 12
  Static physician's global assessment (sPGA) of psoriasis is an average assessment of all psoriatic lesions based on erythema, induration, and scale. It's a 5-point scale performed by investigators. A sPGA score of 0 or 1 means "clear" or "almost clear" respectively.

SECONDARY OUTCOMES:
Incidence, severity and association with the study drug of adverse events (AEs), serious AEs (SAEs), and AEs leading to discontinuation | Baseline to Week 16
Number of participants with clinical laboratory abnormalities | Baseline to Week 16
  Clinical laboratory tests include hematology, coagulation testing, blood chemistry, urinalysis, stool analysis, C-reactive protein, etc.
Incidence of clinically significant changes in electrocardiogram (ECG) | Baseline to Week 16
  ECG parameters include heart rate, PR interval, RR interval, QRS duration, QTcF interval.
Number of participants with abnormalities of physical examination | Baseline to Week 16
  Physical examination includes assessments of general appearance, skin, lymph nodes, head, neck, lung, heart, abdomen, spine, extremities, nervous system, etc.
Number of participants with abnormalities of vital signs | Baseline to Week 16
  Vital signs measured include blood pressure, pulse rate, and temperature.
Proportion of patients with sPGA 0/1 at specified time points | Baseline to Week 16
  Static physician's global assessment (sPGA) of psoriasis is an average assessment of all psoriatic lesions based on erythema, induration, and scale. It's a 5-point scale performed by investigators. A sPGA score of 0 or 1 means "clear" or "almost clear" respectively.
Proportion of patients achieving BSA 75 response at specified time points | Baseline to Week 16
  Psoriasis body surface area (BSA) involvement is measured using the handprint method with the size of a patient's handprint representing ~1% of body surface area involved. BSA 75 response is defined as 75% or greater improvement in BSA score from baseline.
Change from baseline in BSA at specified time points | Baseline to Week 16
  Psoriasis body surface area (BSA) involvement is measured using the handprint method with the size of a patient's handprint representing ~1% of body surface area involved.
Proportion of patients who achieved BSA ≤ 1% at specified time points | Baseline to Week 16
  Psoriasis body surface area (BSA) involvement is measured using the handprint method with the size of a patient's handprint representing ~1% of body surface area involved.
Change from baseline in PASI at specified time points | Baseline to Week 16
  Psoriasis Area and Severity Index (PASI) is a scoring system quantifying the severity of psoriasis based on both lesion severity and area of involvement. PASI assessment is performed by investigators, and the numeric score ranges from 0 to 72, with higher PASI scores denoting more severe disease activity.
Proportion of patients who achieved BSA ≤ 3% for patients with baseline BSA > 3% at specified time points | Baseline to Week 16
  Psoriasis body surface area (BSA) involvement is measured using the handprint method with the size of a patient's handprint representing ~1% of body surface area involved.
Proportion of patients achieving ss-PGA 0/1 for patients with a baseline ss-PGA score ≥2 at specified time points | Baseline to Week 16
  Scalp specific physician's global assessment (sPGA) of psoriasis is an assessment of the disease severity of scalp psoriasis based on erythema, thickness, and scale. It's a 5-point scale performed by investigators. A sPGA score of 0 or 1 means "absence of disease" or "very mild disease" respectively.
Change from baseline in DLQI scores at specified time points | Baseline to Week 16
  The dermatology life quality index (DLQI) is a patient reported outcome measurement. It's a questionnaire consisting of 10 questions concerning patients' perception of the impact of skin diseases on different aspects of their health-related quality of life over the last week. Each question is scored on a scale of 0 to 3, and the sum of each scores range from 0 (no impairment of life quality) to 30 (maximum impairment).

CONTACTS AND LOCATIONS:
Overall Officials: Yuling Shi, MD, Principal Investigator — Shanghai Dermatology Hospital
Locations (1):
- Shanghai Dermatology Hospital, Shanghai, Shanghai Municipality, China